CLINICAL TRIAL: NCT07213024
Title: Social and Physical Activity as Rehabilitation for Preschool Kids With Cancer (SPARK)
Brief Title: Social and Physical Activity as Rehabilitation for Preschool Kids With Cancer
Acronym: SPARK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other); Danish Child Cancer Foundation (Other)
Responsible Party: Principal Investigator, Hanne Baekgaard Larsen, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: p-2024-17472; H-25047770 (Other: Committee on Health Research Ethics, Denmark)
Record Dates: First submitted 2025-10-02; First posted 2025-10-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer; Pediatric Cancer Patients
Keywords: Physical activity; preschool; children; cancer; gross motor function; active play
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: The intervention is a parallel model where the participants are randomized to one of two intervention arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (a) (Experimental): The first intervention arm (a) includes standard care and nine months of facilitated group-structured active play at the hospital. Standard care in-cludes occupational therapy and physiotherapy if needed.
  Interventions: Behavioral: Facilitated group-structured active play at the hospital
- Intervention arm (b) (Experimental): The second intervention arm (b) includes standard care and nine months of facilitated group-structured active play at the hospital combined with a parent educational program and online facilitated structured active play at home. The different intervention components are described in detail below. Standard care includes occupational therapy and physiotherapy if needed.
  Interventions: Behavioral: Facilitated group-structured active play at the hospital; Behavioral: Parents educational program; Behavioral: Online facilitated structured active play at home

INTERVENTIONS:
Behavioral: Facilitated group-structured active play at the hospital — The hospital-based part of the intervention includes daily facilitated group-structured active play sessions during the weekdays (i.e., Monday-Friday) at the hospital for 40 weeks. All sessions will be 45 minutes long and structured using the RePlay Model following four core principles: 1) ritual practices; 2) reinforcement of movement through repetition; 3) devel-opment through appropriate challenges; and 4) adjusting activities to accommodate treat-ment-related side effects. All activities are performed together, where healthcare pro-fessionals, parents, and children all participate to support social development.
  The group-structured active play sessions will take place at the pediatric oncology ward and will be facilitated by a health professional (i.e., an exercise professional or physiother-apist).
Behavioral: Parents educational program — The parent educational program consists of two educational sessions within the first three months of the child's treatment trajectory. The sessions have the aim of providing the par-ents with knowledge and skills to facilitate structured active play at home:
  1. A 30-60-minute session with general information on gross motor function development, common physical side effects of cancer treatment, and the importance of physical activity and active play.
  2. A 60-minute practical, interactive introduction to structured active play and the RePlay Model - including inspiration for active play activities they can do at home that challenge different gross motor skills.
  The parents will receive practical material on gross motor development stages and skills as well as descriptions of active play activities that target gross motor functions.
  Arms: Intervention arm (b)
Behavioral: Online facilitated structured active play at home — The online facilitated structured active play sessions at home are provided daily during the weekdays (i.e., Monday-Friday) in the afternoon (e.g., 16.00-17.00). A healthcare profes-sional (i.e., an exercise professional or physiotherapist) facilitates these sessions, guiding the families through active play activities following the RePlay Model structure. When the families log on for the online sessions, a healthcare professional will instruct them through different play activities. Each family will receive basic essential home-structured active play equipment (e.g., bean bags, balls, bingo games, items for an obstacle course) for the online sessions. The sessions will be conducted through video connections (Teams or Skype). Families who do not have an iPad or suitable computer will receive an iPad from the research group for the nine-month intervention.
  Arms: Intervention arm (b)

SUMMARY:
Physical activity and play in early childhood are positively associated with healthy growth and gross motor, social, and cognitive development. Preschool children with cancer are at risk of impairments or delays in these interdependent developmental areas. Therefore, it is imperative to find new rehabilitation approaches to ensure preschool children's development during and after treatment. This study is based on the RePlay trial, where results highlight a demand from families for physical activity during cancer treatment and show that preschoolers want to participate. However, there is a need for a more flexible and accessible physical activity initiative at the hospital and greater support and collaboration with parents, also at home.

The purpose of this randomized controlled study is to investigate the effect of 9 months of physical activity at the hospital and at home for 82 preschool children with cancer, aged 1-5 years. The rehabilitation program includes the following components:

1. Facilitated structured active play as group sessions at the hospital
2. A parent education program
3. Online facilitated structured active play in the families' homes The included children will be randomized to either a group only receiving structured active play at the hospital (part 1), or a group receiving both structured active play at the hospital, the parent education program, and online structured active play in the families' homes (parts 1-3).

We will measure the children's in gross motor function 9 months after the start of treatment (primary outcome), as well as parents' attitudes towards physical activity and the children's general physical function (secondary outcomes). We will measure at treatment initiation, and 6, 9, and 12 months after treatment initiation. Additionally, we will qualitatively investigate the parents and children's experiences, the potential of the rehabilitation program for the children's social development, and the importance of the professional in facilitating structured active play.

DETAILED DESCRIPTION:
1. BACKGROUND Physical activity and play in early childhood are positively associated with healthy growth and development, this includes motor development (e.g., gross motor functions); psycho-social health (e.g., personal development of self-concept and self-esteem); cognitive de-velopment (e.g., language); and social development (e.g., social skills and functioning). Preschool children diagnosed with cancer are at risk of impairments or delays in several of these interdependent developmental areas. Studies have shown impairments of fine- and gross motor skills during treatment for preschool children with cancer, including severe walking difficulties and loss of ability to support themselves on their legs which limit their movement possibilities and development. Furthermore, these children are taken out of their usual social context in daycare, which limits their social interactions with their peers. When the children re-enter everyday life in daycare, they have trouble following along with their peers physically, have less confidence in their movement abilities, lack age-specific social competencies, and feel excluded. Additionally, one study has shown that these im-pairments persist up to two years after treatment, where the children struggle with develop-ing balance skills and more complex motor skills requirements that come with age. Pre-school children make up half of the population of children who are diagnosed with cancer each year; thus, finding novel rehabilitation approaches to ensure preschoolers' develop-ment during and after cancer treatment is imperative.

   The present trial is based on the experiences within the research group from the RePlay trial (Rehabilitation including structured active play for preschoolers with cancer); the first and largest trial investigating the effect of structured active play as a physical activity inter-vention specifically developed for preschoolers during cancer treatment. The current find-ings highlight a demand from families for physical activity during cancer treatment and show that preschool children want to participate. However, there is a need for a more flexi-ble and easily accessible (i.e., offered all weekdays, located at the ward close to the pa-tients) physical activity intervention at the hospital to increase participation and support the social potential. Furthermore, emphasis is needed on the home-based part of the interven-tion as treatment protocols and isolation requirements have changed so families are more at home during treatment. Preschool children need to be physically active and move as much as possible every day; thus, this calls for an approach with greater support and col-laboration with parents and increased physical activity at home, such as facilitated online physical activity sessions, which have been shown to increase participation in physical activity in older children with cancer.

   Based on our current knowledge and evidence, we have designed Social and Physical Activity as Rehabilitation for preschool Kids with cancer (SPARK)-a randomized con-trolled trial. SPARK includes facilitated group-structured active play at the hospital, based on the RePlay Model, combined with a parent educational program and facilitated online structured active play sessions at home. With this new study, we aim to:
   * Primarily investigate the effect of a nine-month physical activity intervention consisting of group-structured active play at the hospital combined with a parent educational program and online structured active play sessions at home on preschoolers' gross motor function development compared with children only receiving group-structured active play at the hospital.
   * Secondarily investigate the parents' perception of physical activity and the children's general physical function, and qualitatively explore the children's and parents' experiences with the intervention.
2. METHODS

Design:

SPARK is a single-center, two-armed, randomized controlled trial. We will include 82 preschool children newly diagnosed with cancer, aged 1-5 years old.

Additionally, data from the RePlay study's control group will be included to compare to an inactive historical control group.

Following baseline assessment, the children will be randomized to one of two intervention arms. We will stratify by age (<36 months and ≥36 months) and diagnosis (hematological cancers, extra-cranial solid tumors, and tumors in the central nervous system).

Intervention:

The SPARK trial consists of two intervention arms. The first intervention arm (a) includes standard care and nine months of facilitated group-structured active play at the hospital. The second intervention arm (b) includes standard care and nine months of facilitated group-structured active play at the hospital combined with a parent educational program and online facilitated structured active play at home. The different intervention components are described in detail below. Standard care includes occupational therapy and physio-therapy if needed.

* Facilitated group-structured active play at the hospital The hospital-based part of the intervention includes daily facilitated group-structured active play sessions during the weekdays (i.e., Monday-Friday) at the hospital for 40 weeks. All sessions will be 45 minutes long and structured using the RePlay Model following four core principles: 1) ritual practices; 2) reinforcement of movement through repetition; 3) devel-opment through appropriate challenges; and 4) adjusting activities to accommodate treat-ment-related side effects (13). All activities are performed together, where healthcare pro-fessionals, parents, and children all participate to support social development. The RePlay Model, with examples of different active play activities, is illustrated in The group-structured active play sessions will take place at the pediatric oncology ward and will be facilitated by a health professional (i.e., an exercise professional or physiother-apist). Respecting age-specific development, children will be divided into two groups: < 36 months and ≥36 months. Admitted families treated in isolation or otherwise prevented from participating in a group session are offered an individual session in their hospital room fa-cilitated by the healthcare professional.
* Parents educational program

The parent educational program consists of two educational sessions within the first three months of the child's treatment trajectory. The sessions have the aim of providing the par-ents with knowledge and skills to facilitate structured active play at home:

1. A 30-60-minute session with general information on gross motor function development, common physical side effects of cancer treatment, and the importance of physical activity and active play.
2. A 60-minute practical, interactive introduction to structured active play and the RePlay Model - including inspiration for active play activities they can do at home that challenge different gross motor skills.

The parents will receive practical material on gross motor development stages and skills as well as descriptions of active play activities that target gross motor functions. The research group will facilitate interaction with the parents about any questions and barriers they might have with performing structured active play at home.

• Online facilitated structured active play at home The online facilitated structured active play sessions at home are provided daily during the weekdays (i.e., Monday-Friday) in the afternoon (e.g., 16.00-17.00). A healthcare profes-sional (i.e., an exercise professional or physiotherapist) facilitates these sessions, guiding the families through active play activities following the RePlay Model structure. When the families log on for the online sessions, a healthcare professional will instruct them through different play activities. Each family will receive basic essential home-structured active play equipment (e.g., bean bags, balls, bingo games, items for an obstacle course) for the online sessions. The sessions will be conducted through video connections (Teams or Skype). Families who do not have an iPad or suitable computer will receive an iPad from the research group for the nine-month intervention.

Sample size:

The following sample size calculation is based on baseline data from the RePlay study of the gross motor sum of standard scores from PDMS-2. With a mean of 20.03 in gross mo-tor function and a standard deviation of 7.4 (unpublished data from RePlay, n=37), a 25% difference between groups, an alpha level of 0.05 and a power of 80%, we need to include 68 preschool children with cancer. Based on experiences from RePlay, we assume that 20% will be unable to complete the primary outcome at the primary end-point. Therefore, we aim to include 82 preschool children with cancer. Based on the deficiencies observed within two weeks of treatment initiation (baseline score of 20.03 gross motor function), we expect a 25% increase to be obtainable over 9 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children newly diagnosed with cancer or cancer-like benign disorders.
* Children between the ages of ≥12 to <72 months at the time of treatment initiation.
* Children undergoing chemotherapy and/or radiation therapy and/or immuno-therapy at the Department for Pediatrics and Adolescent Medicine at Copenhagen Univer-sity Hospital-Rigshospitalet.

Exclusion Criteria:

* Children diagnosed with severe mental or physical disorders that prevent them from follow-ing instructions in relation to the intervention and testing.
* Children where neither of the parents/guardians can communicate in Danish without a translator.

Ages: 12 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Gross motor function | At treatment initiation (baseline) and 6, 9 (primary end-point), and 12 months (follow-up) after treatment initiation.
  Gross Motor Function is measured with the gross motor function subscale of Peabody Developmental Motor Scales, Third Edition (PDMS-3). PDMS-3 gives a gross motor standard score summed by the standard score from the three gross motor domians; body control, body transport and object control. The primary endpoint is after nine months.

SECONDARY OUTCOMES:
Level of child's function in everyday life | At treatment initiation (baseline) and 6, 9 (primary end-point), and 12 months (follow-up) after treatment initiation.
  Level of function is measured through parent structured interviews with Pediatric Evaluation of Disability Inventory (PEDI) where parents answer wuestions about their child's function in three domains self-care, mobiliy and social functioning and the child's need for help in the same three domains. The primary endpoint is after nine months.
Parents' knowledge | At treatment initiation (baseline), pre and post the parent educational program, and 12 months (follow-up) after treatment initiation.
  We developed a Multiple-Choice Assessment with a one-best-answer format to assess the parent educational program by testing parents' knowledge of physical activity, gross motor development, and structured active play.

OTHER OUTCOMES:
Qualitative explorations | Throughout the intervention and at post intervention at 9 months
  We expect to conduct additional studies that will include empirical data collected through semi-structured interviews and observations. The empirical data collected will be analyzed and reported in separate articles. The children and the parents will be interviewed (parents through semi-structured interviews and children through informal conversations). Observational fieldwork will be carried out during the intervention. The interviews with parents are done during the intervention. The informal conversations and observations are done throughout the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hanne B Larsen, PhD, MSc, RN, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nielsen MKF, Christensen JF, Frandsen TL, Thorsteinsson T, Andersen LB, Christensen KB, Wehner PS, Hasle H, Adamsen LO, Schmiegelow K, Larsen HB. Effects of a physical activity program from diagnosis on cardiorespiratory fitness in children with cancer: a national non-randomized controlled trial. BMC Med. 2020 Jul 6;18(1):175. doi: 10.1186/s12916-020-01634-6. PMID 32624004
- [Background] Stahlhut M, Christensen J, Aadahl M. Applicability and intrarespondent reliability of the pediatric evaluation of disability inventory in a random Danish sample. Pediatr Phys Ther. 2010 Summer;22(2):161-9. doi: 10.1097/PEP.0b013e3181dbf965. PMID 20473099
- [Background] Folio MR, Fewell RR. Peabody Developmental Motor Scales - Second Edition - Examiner's Manual. Second Edi. Austin, TX: PRO-ED; 2000.
- [Background] Keech JJ, Hatzis D, Kavanagh DJ, White KM, Hamilton K. Parents' role constructions for facilitating physical activity-related behaviours in their young children. Aust J Psychol. 2018;70(3):246-57.
- [Background] Trost SG, Loprinzi PD. Parental Influences on Physical Activity Behavior in Children and Adolescents: A Brief Review. Am J Lifestyle Med. 2011;5(2):171-81.
- [Background] Gaser D, Peters C, Oberhoffer-Fritz R, Gotte M, Feuchtinger T, Schmid I, Haller B, von Luettichau I, Kesting S. Effects of strength exercise interventions on activities of daily living, motor performance, and physical activity in children and adolescents with leukemia or non-Hodgkin lymphoma: Results from the randomized controlled ActiveADL Study. Front Pediatr. 2022 Nov 8;10:982996. doi: 10.3389/fped.2022.982996. eCollection 2022. PMID 36425395
- [Background] Thorsteinsson T, Schmiegelow K, Thing LF, Andersen LB, Helms AS, Ingersgaard MV, Lindgren LH, Larsen HB. Classmates motivate childhood cancer patients to participate in physical activity during treatment: A qualitative study. Eur J Cancer Care (Engl). 2019 Sep;28(5):e13121. doi: 10.1111/ecc.13121. Epub 2019 Jun 18. PMID 31215079
- [Background] Pouplier A, Fridh MK, Christensen J, Hoyer A, Schmidt-Andersen P, Winther H, Larsen HB. Rehabilitation including structured active play intervention for preschoolers with cancer during treatment: A RePlay qualitative study of parents' experiences. Eur J Oncol Nurs. 2024 Aug;71:102639. doi: 10.1016/j.ejon.2024.102639. Epub 2024 Jun 7. PMID 38878692
- [Background] Pouplier A, Larsen HB, Christensen J, Schmidt-Andersen P, Winther H, Fridh MK. The rehabilitation including structured active play (RePlay) model: A conceptual model for organizing physical rehabilitation sessions based on structured active play for preschoolers with cancer. Front Pediatr. 2022 Sep 27;10:980257. doi: 10.3389/fped.2022.980257. eCollection 2022. PMID 36238603
- [Background] Pouplier A, Fridh MK, Christensen J, Ruiz-Molsgaard H, Hoyer A, Schmidt-Andersen P, Winther H, Larsen HB. The potential of structured active play for social and personal development in preschoolers during cancer treatment: A qualitative RePlay study. J Adv Nurs. 2024 Apr;80(4):1607-1618. doi: 10.1111/jan.15923. Epub 2023 Nov 10. PMID 37950393
- [Background] Pouplier A, Fridh MK, Schmidt-Andersen P, Nielsen AML, Winther H, Christensen J, Larsen HB. Evaluating the feasibility of a rehabilitation intervention including physical activity as structured active play for preschoolers diagnosed with cancer during the first 6 months of treatment-a study based on data from the RePlay trial. Eur J Pediatr. 2025 Aug 6;184(8):533. doi: 10.1007/s00431-025-06350-y. PMID 40764830
- [Background] Pouplier A, Winther H, Christensen J, Schmidt-Andersen P, Zhang H, Frandsen TL, Schmiegelow K, Fridh MK, Larsen HB. Rehabilitation Including Structured Active Play for Preschoolers With Cancer (RePlay)-Study Protocol for a Randomized Controlled Trial. Front Pediatr. 2022 May 9;10:834512. doi: 10.3389/fped.2022.834512. eCollection 2022. PMID 35615627
- [Background] Darcy L, Enskar K, Bjork M. Young children's experiences of living an everyday life with cancer - A three year interview study. Eur J Oncol Nurs. 2019 Apr;39:1-9. doi: 10.1016/j.ejon.2018.12.007. Epub 2018 Dec 23. PMID 30850132
- [Background] Darcy L, Knutsson S, Huus K, Enskar K. The everyday life of the young child shortly after receiving a cancer diagnosis, from both children's and parent's perspectives. Cancer Nurs. 2014 Nov-Dec;37(6):445-56. doi: 10.1097/NCC.0000000000000114. PMID 24406380
- [Background] De Luca CR, McCarthy M, Galvin J, Green JL, Murphy A, Knight S, Williams J. Gross and fine motor skills in children treated for acute lymphoblastic leukaemia. Dev Neurorehabil. 2013 Jun;16(3):180-7. doi: 10.3109/17518423.2013.771221. Epub 2013 Mar 11. PMID 23477341
- [Background] Vainionpaa L. Clinical neurological findings of children with acute lymphoblastic leukaemia at diagnosis and during treatment. Eur J Pediatr. 1993 Feb;152(2):115-9. doi: 10.1007/BF02072486. PMID 8444217
- [Background] Harman JL, Wise J, Willard VW. Early intervention for infants and toddlers: Applications for pediatric oncology. Pediatr Blood Cancer. 2018 May;65(5):e26921. doi: 10.1002/pbc.26921. Epub 2017 Dec 22. PMID 29271555
- [Background] Carson V, Hunter S, Kuzik N, Wiebe SA, Spence JC, Friedman A, Tremblay MS, Slater L, Hinkley T. Systematic review of physical activity and cognitive development in early childhood. J Sci Med Sport. 2016 Jul;19(7):573-8. doi: 10.1016/j.jsams.2015.07.011. Epub 2015 Jul 10. PMID 26197943
- [Background] Leonard HC, Hill EL. Review: The impact of motor development on typical and atypical social cognition and language: a systematic review. Child Adolesc Ment Health. 2014 Sep;19(3):163-170. doi: 10.1111/camh.12055. Epub 2014 Feb 8. PMID 32878369
- [Background] Timmons BW, Leblanc AG, Carson V, Connor Gorber S, Dillman C, Janssen I, Kho ME, Spence JC, Stearns JA, Tremblay MS. Systematic review of physical activity and health in the early years (aged 0-4 years). Appl Physiol Nutr Metab. 2012 Aug;37(4):773-92. doi: 10.1139/h2012-070. PMID 22765840